CLINICAL TRIAL: NCT03436186
Title: Objective Analysis of Swallowing and Functional Voice Outcomes After Thyroidectomy: A Prospective Cohort Study
Brief Title: Swallowing and Voice Outcomes After Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozer Makay, ass. prof. ozer makay, Ege University
Other Study IDs: tgumus1
Record Dates: First submitted 2018-02-03; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Functional Voice and Swallowing Outcomes
Keywords: Thyroidectomy; voice; swallowing problems; dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- no arm: no arm

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
Impairment in voice and swallowing functions are common after thyroidectomy. The investigators aimed to evaluate the objective functional voice and swallowing outcomes in a series of patients undergoing thyroidectomy.

according to the study, even in the absence of recurrent laryngeal nerve injury, subjective and objective swallowing and voice alterations do occur after thyroidectomy.

DETAILED DESCRIPTION:
A total of 43 consenting patients who underwent thyroidectomy were prospectively recruited. Subjective evaluation of swallowing was assessed with 'Swallowing Impairment Score' and 'MD Anderson Dysphagia Inventory'. Fiberoptic endoscopic evaluation of swallowing (FEES) was applied for objective evaluation. Also, functional oral intake scale (FOIS) and functional outcome swallowing scale (FOSS) were used for swallowing assessment. Voice evaluation was assessed with videostrobolaryngoscopy (VSL) and 'The Multi-Dimensional Voice Program (MDVP)' was used for capturing and analyzing the voice samples. All evaluations were performed preoperatively and on 1st day, 2nd week and 6th months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thyroidectomy

Exclusion Criteria:

* Patients who were diagnosed with thyroid carcinoma preoperatively
* Having history of previous neck surgery,
* History of radiotherapy at head and neck region,
* Vocal cord paralysis,
* neuromuscular dysfunction,
* larynx, esophagus and chest pathology
* who did not want to be involved in the study

Ages: 27 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who underwent thyroidectomy without recurren nerve injury
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
the intake of fluid and thickened liquid food | 6 months
  comparison of the intake of fluid and thickened liquid food between pre- and post-operative scores
light and moderate residual accumulation in solid food intake | 6 months
  comparison of light and moderate residual accumulation in solid food intake between groups
functional oral intake score | 6 months
  comparison of functional oral intake score of specific functional limitation between groups
voice evaluation | 6 months
  comparison of standard deviation of average, fundamental frequency and degree of subharmonics between groups
Swallowing impairment score (SIS) | 6 months
  comparison of Swallowing impairment score (SIS) between pre- and post-operative groups
MD Anderson dysphagia inventory (MDADI) | 6 months
  comparison of MD Anderson dysphagia inventory (MDADI) between pre- and post-operative groups

SECONDARY OUTCOMES:
objective and subjective values correlation | 6 months
  Subjective data showed no correlation with objective findings (p>0.05)

IPD SHARING:
Plan to Share IPD: Undecided
ı dont want to share for 2 years

REFERENCES:
- [Derived] Gumus T, Makay O, Eyigor S, Ozturk K, Erdogan Cetin Z, Sezgin B, Kolcak Z, Icoz G, Akyildiz M. Objective analysis of swallowing and functional voice outcomes after thyroidectomy: A prospective cohort study. Asian J Surg. 2020 Jan;43(1):116-123. doi: 10.1016/j.asjsur.2019.04.013. Epub 2019 May 23. PMID 31130500